CLINICAL TRIAL: NCT04476095
Title: Effects of Photobiomodulation Therapy (PBMT) on Pain Intensity in Patients With Low Back Pain (LBP)
Brief Title: Photobiomodulation Therapy (PBMT) in Patients With Low Back Pain (LBP)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Nove de Julho (Other)
Collaborators: Multi Radiance Medical (Industry); Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Ernesto Cesar Pinto Leal Junior, Full professor, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2.732.044
Record Dates: First submitted 2020-07-09; First posted 2020-07-17 (Actual); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: Low Back Pain
Keywords: Photobiomodulation Therapy
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A researcher will program the device (placebo PBMT or active PMBT) and will be instructed not to inform the patients or other researchers as to the type of treatment (PMBT or placebo). Therefore, the researcher responsible for the treatment, the investigator and the outcome assessor will be blinded to the type of treatment being administered to the patients. The sounds and signals emitted from the device as well as the information displayed on the screen will be identical, regardless of the type of treatment (placebo or PBMT).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Active PBMT (Experimental): Active PBMT will be performed twice a week (at the same time of the day), with intervals of three or four days between sessions, during three-week period (a total of 6 sessions).
  Interventions: Device: Active PBMT
- Placebo PBMT (Placebo Comparator): Placebo PBMT will be performed twice a week (at the same time of the day), with intervals of three or four days between sessions, during three-week period (a total of 6 sessions).
  Interventions: Device: Placebo PBMT

INTERVENTIONS:
Device: Active PBMT — Active PBMT will be applied using a device with 152 emitters (wavelength - 808 nm; dose - 3000 J; treatment time - 600 s), in the low back region.
  Arms: Active PBMT
Device: Placebo PBMT — The placebo PBMT will be applied using the same device as that of active PBMT but without any emission of therapeutic dose. Moreover, the irradiated site and the irradiation time were the same as that of active PBMT. Patients received a total dose of 0 J in the placebo mode. The sounds and signals emitted from the device as well as the information displayed on the screen will be identical, regardless of the type of treatment (active or placebo).
  Arms: Placebo PBMT

SUMMARY:
Low back pain (LBP) is a highly prevalent condition worldwide and the leading cause of years lived with disability. In most cases, the specific pathological cause remains unidentified; therefore, the term non-specific low back pain is commonly used for such cases. Many non-pharmacological therapies are available for the treatment of low back pain aiming to reduce pain and disability. Among these options, photobiomodulation therapy (PBMT) it seems to be an interesting alternative. PBMT is a non-thermal and non-invasive clinical treatment, which has shown effects in decreased pain, modulation of inflammatory process, and tissue repair in musculoskeletal disorders. Therefore, the aim of this project is to evaluate the effects of the PBMT against placebo on pain intensity in patients with chronic non-specific low back pain.

DETAILED DESCRIPTION:
To achieve the proposed objective, it will be performed a randomized, triple-blind (patients, therapists, and outcome assessors), placebo-controlled trial.

Seventy-two patients with chronic non-specific low back pain will be randomly allocated to two treatment groups: 1. Active PBMT or Placebo PBMT.

In both groups, six treatment sessions will be performed twice a week (at the same time of the day), with intervals of three or four days between sessions, during three-week period. The patients will be treated by a blinded therapist.

The outcomes will be obtained at stabilization phase (during 2 weeks), baseline, end of treatment, 24, 48 and 72 hours after the last treatment session, and 7 days after conclusion of treatment. The data will be collected by a blinded assessor.

Statistical analyzis:

* The Fischer's Exact Test will be conducted to compare the proportion of successes between groups.
* The Unpaired t-test will be used for demographic data.
* Repeated measures ANOVA will be performed to analyze pain intensity. The level of statistical significance will be set at p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic non-specific low back pain, with symptoms present for at least three months;
* Patients with a pain intensity of at least 50mm (measured by a 0-100 mm Visual Analog Scale);

Exclusion Criteria:

* Serious spinal pathologies (such as fractures, tumors, inflammatory, and infectious diseases);
* Patients who used local corticosteroids and/or botulin toxin injection for pain relief within the prior 30 days of the beginning of the study;
* Chronic pain diseases as fibromyalgia and diabetic type 1;
* Neuropathic pain;
* Previous spinal surgery in the past 12 months;
* Cancer patients;
* Pregnancy or breast feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2020-07-15 (Estimated); Primary Completion 2020-09-02 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | 3 weeks (end of treatment)
  Pain intensity will be measured by 0-100 standardized Visual Analog Scale (VAS).

SECONDARY OUTCOMES:
Subject satisfaction | 3 weeks (end of treatment).
  Subject satisfaction will be measured by scale uses the following responses: "very satisfied", "somewhat satisfied", "neither satisfied nor dissatisfied", "not very satisfied" or "not at all satisfied".
Control of concomitant medication intake | 3 weeks (end of treatment).
  The control of concomitant medication intake will be measured by a individualized pain management diary.
Pain intensity | 24 hours, 48 hours, and 72 hours after the last treatment session, and 7 days after conclusion of treatment.
  Pain intensity will be measured by 0-100 standardized Visual Analog Scale (VAS).

CONTACTS AND LOCATIONS:
Locations (1):
- Laboratory of Phototherapy and Innovative Technologies in Health, São Paulo, Brazil